CLINICAL TRIAL: NCT03813589
Title: State of congEstive heArt Failure Before the onSet of atrIal Tachyarrhythmias Detected by Implanted devicE in Pacemaker Patients (SEASIDE)
Brief Title: Congestive Heart Failure and Atrial Tachyarrhythmias in Pmk Patients
Acronym: SEASIDE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: San Leonardo Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Russo, MD, San Leonardo Hospital
Other Study IDs: SS001
Record Dates: First submitted 2019-01-20; First posted 2019-01-23 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure，Congestive; Atrial Arrhythmia
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- PMK patients: Patients already implanted with double chamber pacemaker able to detect automatically congestive heart failure and collect atrial events.

SUMMARY:
The aim is to correlate relationship between congestive heart failure and onset of atrial tachyarrhythmias in pacemaker patients. Both atrial events and state of congestive heart failure are collected automatically by implanted device.

ELIGIBILITY:
Inclusion Criteria:

* Recent implant of DR pacemaker according to current guidelines
* Sinus Rhythm at enrollment

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients implanted with dual chamber pacemaker able to automatically detect congestive heart failure and atrial tachyarrhythmias events.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate relationship between atrial tachyarrhythmias and congestive heart failure | twelve months
  Relationship between thoracic impedance variations and atrial events collected by device

SECONDARY OUTCOMES:
Detect optimal device programming | twelve months
  Identify useful index congestion trigger value

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Russo, MD, Principal Investigator — San Leonardo Hospital
Locations (1):
- San Leonardo Hospital, Castellammare di Stabia, Napoli, Italy